CLINICAL TRIAL: NCT06536153
Title: Maternal Under-nutrition and Effect of Amaranth Grain Flat-bread on Anemia in Northern Zone of Sidama Region, Ethiopia.
Brief Title: Maternal Under-nutrition and Effect of Amaranth Grain Flat-bread on Anemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hawassa University (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Amanuel Yoseph Samago, Principal Investigator, Hawassa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB/027/16
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Maternal Anemia in Pregnancy, Before Birth; Maternal; Malnutrition, Affecting Fetus
Keywords: Pregnant women; Undernutrition; Anemia; Amaranth grain; Sidama region; Ethiopia
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Intervention Model Description: Both bi-variable and multivariable analyses using multilevel mixed effects modified Poisson models with random effects will be carried out if the outcome variable prevalence is greater than 20%. If the prevalence is less than 20%, a multilevel mixed effects binary logistic regression model will be utilized to adjust for between- and within-cluster variation for adjusted analysis.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The trial subjects, bread distributors, and outcome assessors (data collectors) will be all unaware of the study groups assignment and bread content. The bread distributers for the maize and amaranth groups will be distinct, and there will be 12 bread-distributers, one for each kebele. Twelve boxes, one for each kebele, will be packed and tagged with the name of the pregnant women. Every day, each bread-distributer fed the pregnant women at their home, under their close supervision. Unopened bread will be returned and recorded by the coordinator each day in the event of absences or refusals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amaranth arm (Experimental): The pregnant women in the experimental group will be referred as the "amaranth arm". Pregnant women in the intervention arm (N = 153) will receive 200 g of flat-bread on a daily basis, comprising 30% chickpea and 70% amaranth grain in mass, for six months.
  Interventions: Combination Product: Amaranth grain flat bread
- Maize arm (Active Comparator): The pregnant women in the control group will be referred as the "maize arm". Pregnant women in the control arm (N = 153) will receive 200 g of bread on a daily basis, comprising 100% maize, for six months.
  Interventions: Combination Product: Amaranth grain flat bread

INTERVENTIONS:
Combination Product: Amaranth grain flat bread — The recipe will be produced according to the recommended dietary allowance (RDA); based on RDA, 200 g of flat-bread (30% chickpea and 70% amaranth grain) comprised 30 mg of iron, which can satisfy 50% of RDA supposing 15-20% iron absorption (54). A prior study concluded that the acceptability was satisfactory in the community (55). Also, a study from the Hawassa University Department of Food Sciences reported that amaranth-grain flat-bread was safe for consumption for 48 hours after preparation and improved the nutritional values (56). To lower the phytate levels in the amaranth grain, home-level processing will be used. For 24 hours, amaranth grain will be soaked in water with 5 milliliters of lemon juice per 100 milliliters of water, and it will germinate for 72 hours. It will be sun-dried, roasted, and ground using a nearby electrical mill before fermented bread is made

SUMMARY:
Introduction: In Ethiopia, maternal malnutrition is a severe public health issue. Underweight and anaemia are the two most common nutritional problems in pregnant women, and they often coexist.

Methods: A community-based cross-sectional study will be undertaken on a sample of 528 pregnant women in their first trimester to investigate the prevalence of anemia and associated risk factors, as well as the prevalence of co-existing anemia and undernutrition. Following that, a six-month parallel-group community-based randomized controlled trial will be conducted among 306 anemic women to assess the effect of locally prepared amaranth grain flatbread on hemoglobin concentration and anemia prevalence when compared to maize bread, which is commonly consumed among pregnant women.

DETAILED DESCRIPTION:
Introduction: In Ethiopia, maternal malnutrition is a major public health concern. Underweight and anaemia are the two most common nutritional disorders in pregnant women, and they frequently co-exist. A prevalent kind of nutritional anaemia is iron-deficiency anaemia (IDA). These issues are primarily caused by a lack of important micro and macronutrients in the diet, as pregnant women eat primarily cereal-based foods. As a result, the burden of under-nutrition in Ethiopia necessitates a more in-depth investigation of underused crops that are high in nutrients and have the potential to minimize food and nutrition insecurity. Although the amaranth plant grows widely in Ethiopia and can boost food intake, its nutritional potential has yet to be acknowledged by community consumers and health professionals.

Methods: A community-based cross-sectional study will be conducted on a sample of 528 pregnant women in their first trimester to examine the prevalence of anemia and identify its risk factors and determine the prevalence of co-existing anemia and under-nutrition among pregnant women. From pregnant women who will be diagnosed for anemia, C-reactive protein (CRP) and serum ferritin will be analyzed to determine IDA. Following this, a parallel-group community-based randomized controlled trial will be conducted for six months among 306 anemic women to evaluate the effect of locally prepared amaranth grain flat-bread on hemoglobin concentration and anemia prevalence compared to the frequently consumed maize bread among pregnant women. A multi-stage sampling method will be utilized to select eligible pregnant women. The households with pregnant women will be identified by conducting the house-to-house census.For categorical variables, summary measures will be presented as absolute frequencies and percentages, but for numerical variables, the mean with standard deviation (SD) will be utilized as a descriptive measure after the distribution is checked for normality. A multi-level mixed-effect logistic/linear regression model will be used to account for between and with cluster effects. We will be used intention-to-treat analyses approach.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women less than 3 months of gestational age and residing in the district for at least 6 months.

Exclusion Criteria:

* Women who have a severe illness during the data collection period
* Women who have a psychiatric disorder
* Women who have plan to change residence during the implementation of an intervention
* Women who have chronic diseases like tuberculosis, HIV/AIDS, and cancer
* women who received blood transfusion in the last 6 months
* Women who have had malaria at least 3 times in the last 3 months
* Women with severe anemia (<7 g/dl) detected during the survey

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 306 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anemia | Up to six months
  In pregnancy, anemia is defined as Hemoglobin <11 g/dl and is classified into three categories based on WHO criteria: mild (10.0-10.9 g/dl), moderate (7.0-9.9 g/dl), and severe (7.0 g/dl)
Prevalence of under-nutrition | Up to six months
  In this study, the MUAC measurements of pregnant mothers who fall below a cutoff point of 23 cm will be classified as undernourished, while those who measure 23 cm or more will be classified as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Amanuel Yo Samago, Masters, Principal Investigator — Hawassa University

IPD SHARING:
Plan to Share IPD: No
SPSS data set will be shared during publication